CLINICAL TRIAL: NCT06995313
Title: Biofeedback Training to Improve Fixation Stability, Visual Function Outcomes, and Quality of Life in Hemianopia Cases
Brief Title: Biofeedback Training for Hemianopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-5618
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hemianopia; Brain Injuries
Keywords: hemianopsia; biofeedback training; brain tumor; brain trauma; visual fields; visual loss; low vision; fixation stability
MeSH Terms: conditions — Hemianopsia; Brain Injuries; Brain Neoplasms; Brain Injuries, Traumatic; Vision Disorders; Vision, Low

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled clinical trial with a treated and a control group without intervention, that will occur in parallel, the control group crossing over to provide additional information.
Who Masked: Outcomes Assessor
Masking Description: The ophthalmic assistants do not have assess to the group the participant is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will receive biofeedback training for 5 weeks in a row, 20 minutes. each session, on the micro perimeter.
  Interventions: Behavioral: Biofeedback training
- Group B (No Intervention): This group will perform the same assessment tests in parallel with Group A and no intervention will be given.

INTERVENTIONS:
Behavioral: Biofeedback training — This is an audio-luminous stimulation on the micro perimeter that teaches the brain to use a different fixation locus on the retinal other than the fovea and develops visual attention to the surrounding retinal areas. 20 minutes exercises for stimulation are performed on the micro perimeter, once a week, for 5 weeks.
  Arms: Group A

SUMMARY:
This is a prospective study that compares biofeedback training on the microperimetry (BT) to a control group in patient s with hemianopia. The patients receive 5 sessions of 20 minutes to stimulate with light and sound the brain in using the best residual area on the visual fields post-brain injury visual loss. Visual tests and quality of life questionnaire are performed pre-and-post-training.

DETAILED DESCRIPTION:
Background

Patients with brain injury secondary to stroke, surgery, or trauma frequently suffer from homonymous hemianopia, defined as vision loss in one hemi-field secondary to retro- chiasma lesion. About 45% of stroke survivors have homonymous hemianopia. A deficit in vision and spatial perception can cause slowdown of the rehabilitation progress in physiotherapy.

Patients face three main visual behavioural problems: (1) impaired eye movements (including saccades) leading to defective visual and spatial exploration, (2) reading deficit ( alexia) because of the para foveal field loss and (3) deviated subjective midline. Dyslexia is not simply the product of the visual field defect but is caused by a disorder of control of visual information processing and eye movements in reading.

Most importantly, the capability to read is fundamental for daily living and an essential prerequisite for education and success in our modern society, so this disorder can have a profound effect on patients' lives. Patients with visual field loss usually fail to adapt to their reading impairment (80% of cases). In these cases, word identification and the abilities to plan and guide reading eye movements are disturbed.

In spite of these facts, visual rehabilitation program on a larger scale is still missing in most rehabilitation centers and clinics. This is decurrent to the generalized belief that lesions of the lateral geniculate nucleus and striate cortex lead to a permanent loss of vision. According to scientific findings, this does not always have to be true.

Optical solutions have shown to be effective in helping visual impairments in hemianopia cases. Relatively small prismatic amounts may be tested and prescribed to this group, as the function of yoked prisms in these cases is to reduce the mismatch between their veridical objective and anomalous subjective sense of straight ahead to a perceptually acceptable level. Yoked prisms have been used by neuro rehabilitative optometrists for decades, as well as others in the field such as occupational therapists, to improve ambulation and gait in hemianopia and/or hemiplegia. Approximately two-thirds of the patients may respond favourably to the yoked prisms. Statements such as 'the visual space seems expanded', and observations such as having improved mobility, ambulation and eye-hand co-ordination, are positive prognostic indicators when prescribing yoked prisms in this diagnostic group.2 Likewise, it was demonstrated that application of yoked prisms improved balance and posture. 'Improved posture, and the sense of feeling more stable while walking through the environment', as well as marked, absence of 'feeling of nausea and dizziness while walking' or 'objects to appear to move when walking'.

Bi temporal visual field impairment frequently leads to binocular vision difficulties. Patients with bi temporal hemianopia with pre-existing strabismus complain of horizontal diplopia, sometimes combined with vertical deviation (with pre-existing). The symptoms are a result of the decompensation into a tropia (slide) due to the lack of retinal correspondence between the remaining nasal fields of both eyes. Aligning the eyes with prisms can prevent diplopia if the bi temporal hemianopia is incomplete.

Classic and effective saccadic compensatory training therapies are current. They aim to reorganize the control of visual information processing and eye movements or, in other words, to induce or improve oculomotor adaptation to visual field loss. Such therapies involve the systematic and repetitive practice of specific eye movements for reading or for visual exploration. Patients learn to intentionally shift their eyes and, thus, their visual field border, into the area corresponding to their blind visual field. This shift brings the visual information from the blind field into the seeing field for further processing. Patients learn, therefore, to efficiently use their eyes "to keep the 'blind side' in sight". The training-induced, efficient oculomotor adaptation to visual field loss becomes manifest as a change of reading (or visual exploration) eye-movement patterns and indicates the functional reorganization of the control of visual information processing and eye movements.

Biofeedback training for active eye movement control was never used in hemianopia cases before. Biofeedback training (BT) is the latest and newest technique for oculomotor control training in cases with low vision when using available modules in the new instruments. Studies in the literature highlighted positive benefits from using BT in a variety of central vision loss, nystagmus cases, and others. The purpose of this study is to assess systematically the impact of BT in a series of cases with hemianopia and formulate guidelines for further use of this intervention in vision rehabilitation of hemianopia cases in general.

Rationale for the study

The deviation of the subjective midline in hemianopia cases brings visual perception from a line of objects in the surrounds to be at a much higher-level of perception/cognition, thus disturbing reading, gait and balance. Besides that, impaired saccades also cause wrong exploration patterns and deteriorated visual search. It results in the prolonged exploration time of a scene and can lead to significant problems in daily life such as inability to navigate around various obstacles (cars, people and other objects). It also causes a cognitive deficit while extracting information from a visual scene. A combination of factors such as reduced contrast sensitivity, impaired visual search and inaccurate fixation contributes to the matter.

Visual information extraction from the para foveal visual field provides the basis for planning and guiding of reading eye movements. Therefore, patients with hemianopia have difficulties in shifting their gaze systematically from left to right (in right-sided field loss) or finding the beginning of a new line (in left sided field loss). Such eye movements are optimized by visual feedback. BT promotes luminous and auditory biofeedback, which increases its efficacy in vision rehabilitation.

BT provides the accurate and efficient oculomotor training necessary to relocate the subjective midline to the seeing field in 1 or even more, as needed. BT also improves dramatically fixation stability and saccades. The advantage of this training method over classic training is potentially great. Firstly, the highest retinal sensitivity convenient point can be identified considering the whole visual field. The device provides real time scrutiny of ocular movements on a screen, and the therapist is able to select precisely the trained retinal locus (FFT) to be used by the patient on top of the visual field. Finally, according to the patients' response the FFT can be readjusted. Eight cases trained with BT for hemianopia in our low vision rehabilitation (LVR) service had marked improvements in fixation stability, and micro perimeter fields.

Expansion of visual space in the direction of the blind field and compression of visual space in the direction of the seeing field may be a contributory factor to the altered perception of their egocentric directional sense and overall more veridical mapping of their visual space, as well as the resultant shift in their positional centre of gravity. We hypothesize that BT promotes this field relocation.

Conventional visual exploration training studies have confirmed that 10 to 25 training sessions in a 6-week period can be effective for hemianopia patients to adopt these strategies. BT is able to achieve significant results in 5 weekly sessions of 20 minutes each, according to 8 cases treated in our service.

Study hypothesis

The visual and audio parts of the BT program improve in a synergistic way oculomotor control through attention improvement and volitional eye movements towards pre-designated targets. Improved oculomotor control results in better fixation stability of eyes. Better fixation stability in turn results in better navigation for distance and near vision reading. Dual sensory BT is a therapy used in low vision for more than ten years, showing good results for near and distance vision in cases with macular degeneration and other pathologies. The study hypothesis, never tested before, is that BT in cases with hemianopia will positively impact oculomotor control and visual acuity as it was proven to do in cases with macular degeneration.

Significance of the study

Vision is a major sensory input to the human brain. Half of the afferent neuronal axons projecting to the brain originate from the eyes. Intact visual abilities are an important condition enabling us to orient ourselves in our world. It was reported that 50% of all neurological admissions into hospitals in the United Kingdom are due to a stroke and 30% percent of them are reported to have hemianopia.

Numbers of patients reported in the Czech Republic are similar and somewhat lower due to differences in diagnostics and classification of nosological units. Visual impairments are present in 20 to 40% of patients in neurological rehabilitation centres.

If brain visual plasticity is possible to be achieved from conventional vision training methods, specialized training with BT needs to be investigated as a tool for improving a cortical visual disorder. There is a need for simple and more effective visual training which could be used in LVR in large scale for hemianopia cases. Furthermore, BT needs to be evaluated in terms of quality of life (QoL) improvement to the patients.

Clinical trial design

This is a prospective clinical randomized trial to include a control group and take place over a period of up to 24 months. 35 patients will be randomized to the treated group (BT) and 35 patients to the control group.

The objectives set for this trial is to verify if BT impacts on oculomotor control in cases with hemianopia and results in better fixation stability, reading speed and QoL in those trained with BT.

Primary endpoints selected for this trial are retinal sensitivity, fixation stability (FS) estimates as tested with the Micro perimetry, Humphrey Full Field 120 perimetry (Carl Zeiss, Germany), reading speed as tested with the reading speed test, and QoL assessed with the 48 questions LVR questionnaire.

Secondary endpoints are preferred retinal locus (PRL) topographic coordinates, as tested with the Micro perimeter, contrast sensitivity measured with the charts, and Best Corrected Visual Acuity (BCVA) scores for distance and near vision tested with ETDRS charts at 4 meters and 33 cm.

Clinical trial population:

The intended population for this clinical trial is to be found among our own practice patients or among patients referred to our low vision rehabilitation practice. We will consider inclusion into the trial patients that meet the trial entry criteria defined below.

Inclusion criteria: hemianopia cases with more than 6 months from the date of the lesion, previously diagnosed accordingly by micro perimetry and other tests as needed, 18-90 years old, ability to follow the visual and auditory stimuli and training instructions.

Exclusion criteria: previous or current treatment for low vision rehabilitation, ocular diseases, other serious clinical conditions not related to the hemianopia, both eyes with media opacity that impairs micro perimetry testing, lack of ability to perform the tests and training.

Clinical trial procedures All parties involved in the conduct of this clinical trial will be qualified by education, training, or experience to perform their tasks, and this training will be documented appropriately. The investigation will not commence after receiving written approval from the ethics board of the University Health Network. All trial staff will be required to undergo training prior to performing any trial-related activities.

The following is an overview of the study procedures: following obtaining consent from study participants, confirmation of eligibility, and baseline visit assessments, patients will be randomized in 2 groups: BT and control. Treated group participants will undergo 5 BT sessions. 30 days after completion of the 5 BT sessions, participants will return for the first follow up visit, followed by follow up visits at 6 months and 1 year post-BT. The control group of participants in the randomized arm will perform the same tests as in the baseline visit at 30 days post-BT and end the participation in the study. After that, the control group will be provided the option to perform the 5 BT sessions. Following completion of the study visits, participants will return to regular clinical care, that includes BT when needed.

The following is a detailed description of the study procedures:

Screening The following information will be evaluated from medical records and documented, to ensure each subject meets entry criteria prior to consent: diagnosis, age, visual impairment, disabilities related to visual impairments and impact of disabilities on quality of life.

Informed consent Informed Consent Forms will be utilized detailing requirements and considerations for patient consent or legal representative. An authorized designee will conduct the informed consent process. This process will include a verbal discussion with the patient / legal representative on all aspects of the clinical trial that are relevant to the participant's decision to participate such as details of the procedures, anticipated benefits, and potential risks of clinical trial participation. During the discussion, the authorized designee will avoid any improper influence on the subject and will respect the subject's legal rights. The patient / representative will be provided with Informed Consent Form approved by the ethics board and written in a language that is understandable to the patient / representative. The participant will have adequate time to review, ask questions and consider participation. If the patient agrees to participate, the Informed Consent Forms will be signed and dated by the patient / legal representative and by the person obtaining the consent. The signed original will be filed in the subject's research charts, and copies will be provided to the participant.

Standard of care procedures: All clinical trial procedures described below are part of the standard of care procedures experienced by patients with the exception of randomization and the following procedure used in the control group: The procedure involves presentation of a standard fixation target (FT) consisting of a small red circle of about 0.76° diameter. Initially the participant will be instructed to stare at the FT circle. Following this stage, the participant will be guided to look at the FT and simultaneously to be aware of any flashing lights in the periphery of vision. As performing this task, the participant will actively control the eye movements and similar to computer games, the patient has to identify targets in the peripheral field of vision and respond by pressing a button.

Baseline procedures

Visit 1: If the patient accepts to take part in this study and signs the consent form, there will be a low vision baseline assessment. This may take about 1 hour. At the time the patient books this assessment, all the procedures for coronavirus screening will be done normally by phone. Before the patient enters the clinic, the screening questions will be repeated, and they should wear a mask all the time during the consultation. Hands hygiene will be facilitated all the way in the clinic, and all the equipment, charts and surfaces will be disinfected pre- and post- examinations. Demographics and medical history will be collected at this time.

During the baseline visit (Visit 1) participants will be assessed for Best Corrected Visual Acuity (BCVA) for distance vision with ETDRS charts at 4 meters, retinal sensitivity and fixation stability (FS) estimates from micro perimetry C 10-2 with the micro perimeter, Perimetry with the Humphrey perimeter (Carl Zeiss, Germany) , and eye movement scanning with the right eye device (pupil tracker). Participants will be assessed also for near vision with the 100% chart and contrast sensitivity measured with the chart. Quality of Life estimates will be assessed with the 48 questions questionnaire. This visit may take up to an hour in total.

Randomization Following the baseline assessment participants will then be randomized in a ratio 1:1 between BT Treatment and Control groups. For this purpose, we will use for all study participants one of the freely available Clinical Trial Randomization Tools by The National Cancer Institute's Division of Cancer Prevention randomization generator.

Study participants will be randomized to:

* Group A (Treatment with BT) will receive the audio biofeedback training and follow up visits at 9 weeks, 6 months, 12 months, and 24 months after baseline visit.
* Group B (Control) will perform a follow up visit at 9 weeks, 6 months, 12 months, and 24 months after baseline visit.

Training procedure BT will take place during a 20 minutes weekly visit to the office. During training procedure visits (Visits 2-6) the participant is seated in front of the instrument. The procedure involves presentation of a standard fixation target (FT) consisting of a small red circle of about 0.76° diameter. A fixation training target (FTT) will be selected by the trainer at a perceived better fixation point. Initially the participant will be instructed to stare at the FT circle. Following this stage, the participant will be guided to look in the direction of the FTT and listen simultaneously to the audio feedback. As performing this task, the participant will actively control the eye movements until the audio feedback becomes more frequent and then becomes a continuous sound pattern. This continuous sound will signalize to the patient that the FTT location was reached.

End of study procedures The final follow up Visit 7 visit will take place at 45 days following visit 6. This visit may take an hour time. At visit 7, repeat assessments will take place for Best Corrected Visual Acuity (BCVA) for distance vision with ETDRS charts at 4 meters, preferred retinal locus (PRL) characteristics, retinal sensitivity and fixation stability (FS) estimates with the micro perimeter. Participants will be assessed also for near vision, reading speed and contrast sensitivity measured with the contrast charts, stereopsis will be assessed with the Stereo Test, and Quality of Life estimates will be assessed with the 48 question questionnaire. After the participation in the study, the patients will continue to be followed in the regular LVR clinic at the same service.

Follow-up duration

Following the completion of biofeedback treatment visits, patients will be followed for 6 months since their initial recruitment for the primary study time-point. Additionally, patients will be followed for up to 2 years for long-term outcomes of the biofeedback treatment. Visits 8, 9 and 10 will follow the same procedures as visit 7 for assessments.

ELIGIBILITY:
Inclusion Criteria:

Hemianopia cases with more than 6 months from the date of the lesion, previously diagnosed accordingly by micro perimetry and other tests as needed, 18-90 years old, ability to follow the visual and auditory stimuli and training instructions.

Exclusion Criteria:

Previous or current treatment for low vision rehabilitation, ocular diseases, other serious clinical conditions not related to the hemianopia, both eyes with media opacity that impairs microperimetry testing, lack of ability to perform the tests and training.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Retinal sensitivity | Pre- intervention and 1 month post-intervention.
  Micro perimeter retinal sensitivity after performing the C 10-2 68 points test.

SECONDARY OUTCOMES:
Quality of Life Self Referred Score | Pre- intervention and 1 month post-intervention.
  Measured by the 48 questions self-referred questionnaire.
Reading Speed | Pre- intervention and 1 month post-intervention.
  Number of words read per minute as measured by the Minnesota App.
Humphrey Perimetry | Pre- intervention and 1 month post-intervention.
  Full Field 120 monocular and Binocular Tests
Best corrected visual acuity for distance and near | Pre- intervention and 1 month post-intervention.
  ETDRS measured
Fixation stability | Pre- intervention and 1 month post-intervention.
  Measured by the micro perimeter for 20 seconds fixating at a single target.
Oculomotor function | Pre- intervention and 1 month post-intervention.
  Measured by the right eye device for circular, horizontal, vertical pursuit, saccades, and fixation

CONTACTS AND LOCATIONS:
Overall Officials: MONICA Daibert Nido, Assistant, Principal Investigator — University Healt Network
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada